CLINICAL TRIAL: NCT04182191
Title: Influence of Cytochrome P450 (CYP2C9) Genotype on Clinical Efficacy of Tenoxicam After Lower Third Molars Surgeries
Brief Title: Influence of CYP2C9 Genotype on Clinical Efficacy of Tenoxicam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Paulo Zupelari Goncalves, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 66699717.3.3001.5417
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Molar, Third; Pain
MeSH Terms: conditions — Pain | interventions — tenoxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional group (Experimental): 89 patients will be treated with tenoxicam (20 mg once daily for 4 days) for pain control after lower third molar surgery
  Interventions: Drug: Tenoxicam

INTERVENTIONS:
Drug: Tenoxicam — After extraction of at least one third molar, 89 patients will be treated with tenoxicam (20 mg once daily for 4 days) for pain control, collect the saliva to be genotyped and phenotyped for CYP2C9 (by PCR) and their post-operative notes (pain, swelling, trismus, temperature) will be analyzed.

SUMMARY:
The goal of this study is to evaluate the different gene haplotypes for the clinical efficacy of tenoxicam after third lower molar surgery for pain, edema and trismus, adverse reactions, need of rescue medication, patient satisfaction regarding the drug and the pharmacokinetics of the drug between the different gene haplotypes for CYP2C9 that are found in this population

DETAILED DESCRIPTION:
Pharmacogenetics is an area of Pharmacology that studies the contribution of genetic factors to individual responses to drugs. This branch of science involves the variability in pharmacodynamics and pharmacokinetics through the study of polymorphisms in genes encoding receptors, as well as in drug metabolism, where this area of Pharmacology has been growing and achieving its first results with clinical use. The NSAIDS are metabolized by cytochrome P450 (CYP) family, predominantly CYP2C9. The goal of this study is to evaluate the different gene haplotypes for the clinical efficacy of tenoxicam after third lower molar surgery for pain, edema and trismus, adverse reactions, need of rescue medication, patient satisfaction regarding the drug and the pharmacokinetics of the drug between the different gene haplotypes for CYP2C9 that are found in this population. Therefore, 100 patients will be genotyped and phenotyped for this gene and their postoperative data will be confronted with the data found in the Brazilian population. For the analysis of the proposed gene, saliva will be collected and serve as a source of genomic DNA. For the molecular analysis, polymerase chain reaction (PCR) with tests validated and produced by Applied Biosystems® will be performed. The analysis of the results will be described with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Impacted lower third molar;
* not making use of nonsteroidal anti-inflammatory drugs in the last 7 days;

Exclusion Criteria:

* Local anesthetics allergy;
* History of gastrointestinal bleeding or ulcers;
* Kidney disease;
* Asthma;
* Allergy or sensitivity to aspirin or any other anti-inflammatory non-steroid agent;
* Pregnant or nursing women;
* Patients using antidepressant, diuretic or aspirin;
* Patients received antibiotics for 30 days prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change of pain measured by visual analogue scale on periods of 0, 025, 05, 0,75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours after surgery. | Three days after surgery
  Change of pain after third molar surgery is measured by visual analogue scale. It is expected that the visual analogue scale 100mm present lower values in patients heterozygous and mutated for the CYP2C9 the evaluated periods of 0, 15, 30,45 min, 1, 2, 3, 4, 5, 6, 8, 12, 16 , 24 48 and 72 hours after surgery. Lower values on this scale means lower pain suffered by the volunteers.

SECONDARY OUTCOMES:
Adverse effects | Seven days after surgery
  Changes on reporting of adverse effects during the postoperative period until suture removal seven days after extraction of third molar included and/or impacted in patients heterozygous or mutated for CYP2C9 assessed by the information contained in the medical records of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Zupelari Goncalves, DDS, Ms, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No